CLINICAL TRIAL: NCT00003025
Title: A Phase I Pilot Trial of Immunotherapy With Autologous Tumor-Derived gp96 Heat Shock Protein - Peptide Complex (HSPPC-96) in Patients With Resected Pancreatic Adenocarcinoma
Brief Title: Vaccine Therapy in Treating Patients With Stage I or Stage II Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 97-034; CDR0000065613 (Registry Identifier: PDQ (Physician Data Query)); ANTIGENICS-C-100-01; NCI-G97-1271
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — vitespin

INTERVENTIONS:
Biological: vitespen

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an immune response to and kill tumor cells. Combining vaccine therapy with surgery may be an effective treatment for pancreatic cancer.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients with stage I or stage II pancreatic cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Study the safety of autologous tumor derived gp96 heat shock protein peptide complex (HSPPC-96) in patients with resected pancreatic adenocarcinoma. II. Examine the immune response to HSPPC-96 in this group of patients.

OUTLINE: This is a dose escalation study. Six weeks after surgery patients are given autologous tumor derived gp96 heat shock protein peptide complex (HSPPC-96) subcutaneously once a week for 4 weeks. Five patients are initially enrolled at each of two dose levels. An additional three patients may be enrolled at each dose level to determine the optimal dose of HSPPC-96. Patients are followed at weeks 1, 4, and 12 after treatment.

PROJECTED ACCRUAL: A maximum of 16 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, resected, stage I or II pancreatic adenocarcinoma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3000/mm3 Lymphocyte count at least 700/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No clinically significant heart disease Other: No other serious illness No active infections requiring antibiotics within past 2 weeks Not pregnant or nursing Fertile patients must use effective birth control No known immunodeficiency No active bleeding

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: No concurrent corticosteroids Radiotherapy: No prior radiation therapy Surgery: Must undergo Whipple procedure or distal pancreatectomy at Memorial Hospital Must not have undergone splenectomy Other: No investigational treatment within 2 months of surgery No immunosuppressive therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 1997-03; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, PhD, FACS, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Maki RG, Lewis JJ, Janetzki S, et al.: Phase I study of HSPPC-96 (oncophage®) vaccine in patients with completely resected pancreatic adenocarcinoma. [Abstract] European Journal of Cancer Supplements 1 (5): A-48, S19, 2003.